CLINICAL TRIAL: NCT02201628
Title: Comparison of Nasopharyngeal and Lower Oesophageal Temperatures Under General Anaesthesia With an Endotracheal Tube With Leak
Brief Title: Correlation of Nasopharyngeal (NP) and Lower Oesophageal (LO) Temperatures in Ventilated Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14SG04
Record Dates: First submitted 2014-07-15; First posted 2014-07-28 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Child
Keywords: Oesophageal; Nasopharyngeal; temperature; Intubation, endotracheal; Pediatric; Anesthesia; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nasopharyngeal and oesophageal temperatures (Experimental): An oesophageal and nasopharyngeal temperature probe will be placed and temperature will be measured at these site
  Interventions: Device: Nasopharyngeal and oesophageal temperature probes

INTERVENTIONS:
Device: Nasopharyngeal and oesophageal temperature probes
  Other Names: Covidien; Mon-a-therm™ General Purpose Temperature Probe 400TM; 90050

SUMMARY:
Children lose heat under general anaesthesia, thus temperature is routinely monitored during anaesthesia for all but the shortest cases, and active warming can be used to prevent hypothermia and its resulting complications. Temperature can be measured at several sites dependent on the type of surgery and patient factors. Previously a temperature probe has been sited in the lower third of the oesophagus (swallowing tube) but it is difficult to accurately place this without an X-Ray. Consequently it is more common to use a temperature probe placed in the nasopharynx (where the nose and throat meet), when the child is anaesthetised.

However the investigators do not know if the temperature in the nasopharynx correlates well with the real core temperature or not.This prospective, unblinded, agreement study will seek to find an agreement of 2 methods to measure temperature in children undergoing general anaesthesia with a breathing tube that has a leak.

DETAILED DESCRIPTION:
It is known that temperature in the lower third of the oesophagus correlates well with the gold standard of core temperature measurement, namely the temperature of blood in the heart. It is not known if oesophageal and nasopharyngeal temperatures correlate in children on a breathing machine via a tube with leak. If this study were to find a good correlation between oesophageal and nasopharyngeal temperature, this would allow clinicians to confidently use the more feasible nasopharyngeal temperature probes.

For this study 100 children will have both nasopharyngeal and oesophageal temperatures measured during general anaesthesia, both in the presence and absence of a leak around the endotracheal tube.

It is hypothesised that even in the presence of a leak, the temperature difference between the two methods will be less than 0.5 degrees centigrade.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires general anaesthesia with endotracheal intubation for a procedure assisted by radiography (e.g. line insertion, line change).
* Patient requires chest radiograph for procedure.
* Expected anaesthetic time more than 30 minutes.

Exclusion Criteria:

* No written parental written consent.
* Known oesophageal pathology (e.g. tracheo-oesophageal fistula, oesophageal strictures, oesophageal varices, oesophageal atresia).
* Known base of skull or midface fractures.
* Previous gastric bypass surgery or nasal surgery.
* Known coagulopathy.
* Previous alkaline ingestion.
* High aspiration risk.
* Significant respiratory co-morbidity requiring anticipated peak airway pressures > 25 cm of water
* American Society Anaesthesiologists (ASA) grading 4 - 5.
* Tracheostomy in situ.
* Severe sepsis or septic shock or other other condition (such as bronchopulmonary fistula) that precludes use of tidal volume ventilation over 7 ml/kg.
* Known airway abnormalities (e.g. subglottic stenosis) that preclude placement of a MicroCuff® endotracheal tube.
* Oesophageal or nasopharyngeal probe contraindicated for reasons related to surgery / procedure.

Ages: 8 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2014-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarjan P Snoek, MBChB, FRCA, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Helen V Hume-Smith, MBBS, FRCA, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Emily Haberman, MBBS, FRCA, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Torossian A. Thermal management during anaesthesia and thermoregulation standards for the prevention of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):659-68. doi: 10.1016/j.bpa.2008.07.006. PMID 19137809
- [Background] Sessler DI. Complications and treatment of mild hypothermia. Anesthesiology. 2001 Aug;95(2):531-43. doi: 10.1097/00000542-200108000-00040. No abstract available. PMID 11506130
- [Background] Evans DC, Doraiswamy VA, Prosciak MP, Silviera M, Seamon MJ, Rodriguez Funes V, Cipolla J, Wang CF, Kavuturu S, Torigian DA, Cook CH, Lindsey DE, Steinberg SM, Stawicki SP. Complications associated with pulmonary artery catheters: a comprehensive clinical review. Scand J Surg. 2009;98(4):199-208. doi: 10.1177/145749690909800402. PMID 20218415
- [Background] Robinson JL, Seal RF, Spady DW, Joffres MR. Comparison of esophageal, rectal, axillary, bladder, tympanic, and pulmonary artery temperatures in children. J Pediatr. 1998 Oct;133(4):553-6. doi: 10.1016/s0022-3476(98)70067-8. PMID 9787697
- [Background] SEVERINGHAUS JW, STUPFEL M. Internal body temperature gradients during anesthesia and hypothermia and effect of vagotomy. J Appl Physiol. 1956 Nov;9(3):380-6. doi: 10.1152/jappl.1956.9.3.380. No abstract available. PMID 13376459
- [Background] Whitby JD, Dunkin LJ. Temperature differences in the oesophagus. Preliminary study. Br J Anaesth. 1968 Dec;40(12):991-5. doi: 10.1093/bja/40.12.991. No abstract available. PMID 5710916
- [Background] Whitby JD, Dunkin LJ. Oesophageal temperature differences in children. Br J Anaesth. 1970 Nov;42(11):1013-5. doi: 10.1093/bja/42.11.1013. No abstract available. PMID 5488350
- [Background] Kaukuntla H, Harrington D, Bilkoo I, Clutton-Brock T, Jones T, Bonser RS. Temperature monitoring during cardiopulmonary bypass--do we undercool or overheat the brain? Eur J Cardiothorac Surg. 2004 Sep;26(3):580-5. doi: 10.1016/j.ejcts.2004.05.004. PMID 15302054
- [Background] Holtzclaw BJ. Monitoring body temperature. AACN Clin Issues Crit Care Nurs. 1993 Feb;4(1):44-55. PMID 8452743
- [Background] Stone JG, Young WL, Smith CR, Solomon RA, Wald A, Ostapkovich N, Shrebnick DB. Do standard monitoring sites reflect true brain temperature when profound hypothermia is rapidly induced and reversed? Anesthesiology. 1995 Feb;82(2):344-51. doi: 10.1097/00000542-199502000-00004. PMID 7856892
- [Background] Maxton FJ, Justin L, Gillies D. Estimating core temperature in infants and children after cardiac surgery: a comparison of six methods. J Adv Nurs. 2004 Jan;45(2):214-22. doi: 10.1046/j.1365-2648.2003.02883.x. PMID 14706007
- [Background] Whitby JD, Dunkin LJ. Cerebral, oesophageal and nasopharyngeal temperatures. Br J Anaesth. 1971 Jul;43(7):673-6. doi: 10.1093/bja/43.7.673. No abstract available. PMID 5564234
- [Background] Litman RS, Maxwell LG. Cuffed versus uncuffed endotracheal tubes in pediatric anesthesia: the debate should finally end. Anesthesiology. 2013 Mar;118(3):500-1. doi: 10.1097/ALN.0b013e318282cc8f. No abstract available. PMID 23314108
- [Background] Strobel CT, Byrne WJ, Ament ME, Euler AR. Correlation of esophageal lengths in children with height: application to the Tuttle test without prior esophageal manometry. J Pediatr. 1979 Jan;94(1):81-4. doi: 10.1016/s0022-3476(79)80361-3. No abstract available. PMID 758430
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Ramsay JG, Ralley FE, Whalley DG, DelliColli P, Wynands JE. Site of temperature monitoring and prediction of afterdrop after open heart surgery. Can Anaesth Soc J. 1985 Nov;32(6):607-12. doi: 10.1007/BF03011406. PMID 3878219
- [Background] Cronin K, Wallis M. Temperature taking in the ICU: which route is best? Aust Crit Care. 2000 May;13(2):59-64. doi: 10.1016/s1036-7314(00)70623-0. PMID 11235453
- [Background] Ko HK, Flemmer A, Haberl C, Simbruner G. Methodological investigation of measuring nasopharyngeal temperature as noninvasive brain temperature analogue in the neonate. Intensive Care Med. 2001 Apr;27(4):736-42. doi: 10.1007/s001340000829. PMID 11398702
- [Background] Muravchick S. Deep body thermometry during general anesthesia. Anesthesiology. 1983 Mar;58(3):271-5. doi: 10.1097/00000542-198303000-00014. No abstract available. PMID 6829963
- [Background] Wass CT, Long TR, Deschamps C. Entrapment of a nasopharyngeal temperature probe: an unusual complication during an apparently uneventful elective revision laparoscopic Nissen fundoplication. Dis Esophagus. 2010 Jan;23(1):33-5. doi: 10.1111/j.1442-2050.2009.00968.x. Epub 2009 Apr 15. PMID 19392849
- [Background] Williams DJ, Kelleher AA. Defective nasopharyngeal temperature probes. Anaesthesia. 2002 Dec;57(12):1223; author reply 1223-4. doi: 10.1046/j.1365-2044.2002.02913_18.x. No abstract available. PMID 12437729
- [Background] Paik UH, Lee TR, Kang MJ, Shin TG, Sim MS, Jo IJ, Song KJ, Jeong YK. Success rates and procedure times of oesophageal temperature probe insertion for therapeutic hypothermia treatment of cardiac arrest according to insertion methods in the emergency department. Emerg Med J. 2013 Nov;30(11):896-900. doi: 10.1136/emermed-2012-201579. Epub 2012 Nov 17. PMID 23161807
- [Background] Smith JH, Keltie K, Murphy T, Raj N, Lane M, Ranger M, Sims AJ. A comparison of three methods that assess tracheal tube leakage: leak conductance, fractional volume loss, and audible assessment. Paediatr Anaesth. 2013 Feb;23(2):111-6. doi: 10.1111/pan.12043. Epub 2012 Oct 13. PMID 23061742
- [Result] Whitby JD, Dunkin LJ. Temperature differences in the oesophagus. The effects of intubation and ventilation. Br J Anaesth. 1969 Jul;41(7):615-8. doi: 10.1093/bja/41.7.615. No abstract available. PMID 5798841
- [Result] Bloch EC, Ginsberg B, Binner RA Jr. The esophageal temperature gradient in anesthetized children. J Clin Monit. 1993 Apr;9(2):73-7. doi: 10.1007/BF01616917. PMID 8478651
- [Result] Mekjavic IB, Rempel ME. Determination of esophageal probe insertion length based on standing and sitting height. J Appl Physiol (1985). 1990 Jul;69(1):376-9. doi: 10.1152/jappl.1990.69.1.376. PMID 2394660
- [Result] Taylor C, Subaiya L, Corsino D. Pediatric cuffed endotracheal tubes: an evolution of care. Ochsner J. 2011 Spring;11(1):52-6. PMID 21603336
- [Result] Matsukawa T, Ozaki M, Sessler DI, Nishiyama T, Imamura M, Kumazawa T. Accuracy and precision of "deep sternal" and tracheal temperatures at high- and low-fresh-gas flows. Br J Anaesth. 1998 Aug;81(2):171-5. doi: 10.1093/bja/81.2.171. PMID 9813517
- [Result] Weiss M, Dullenkopf A, Fischer JE, Keller C, Gerber AC; European Paediatric Endotracheal Intubation Study Group. Prospective randomized controlled multi-centre trial of cuffed or uncuffed endotracheal tubes in small children. Br J Anaesth. 2009 Dec;103(6):867-73. doi: 10.1093/bja/aep290. Epub 2009 Nov 3. PMID 19887533
- See also: National Institute for Health and Clinical Excellence. The management of inadvertent perioperative hypothermia in adults: full guideline — https://www.nice.org.uk/guidance/cg65/update/CG65/documents/perioperative-hypothermia-inadvertent-guideline-full-guideline-part-12

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 were excluded due to incomplete data or insufficient FVL difference between cuff down and cuff up scenarios
Groups:
- Cuff Inflation and Cuff Deflation Groups: Cuff deflation to achieve softly audible leak. Cuff inflation means no leak or minimal leak
Period: Overall Study
Arm/Group | Cuff Inflation and Cuff Deflation Groups
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cuff Inflation and Cuff Deflation Groups
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.3 [1.8 to 5.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50

OUTCOME MEASURES:

1. Primary Outcome: Temperature Difference (in Degrees Celsius) Between 2 Body Sites in Children Undergoing General Anaesthesia. The 2 Sites Are: (1) Lower Oesophagus; (2) Nasopharynx
Description: Temperature will be measured in the lower oesophagus of a child ventilated with a cuffed Endotracheal Tube (ETT). Readings will be recorded when there is no leak (cuff up) and when there is a clinically determinable, soft, audible leak (cuff down) around the ETT. Simultaneously temperature will also be measured in the nasopharynx.
  This will occur during general anaesthesia for a procedure that entails the performance of a radiograph (X-Ray) of the chest. The X-Ray will be used by the investigators to confirm correct placement of the temperature probe in the lower third of the oesophagus. We aim to show that the temperature measured in the lower oesophagus is the same or does not significantly differ from the temperature in the nasopharynx, even in the presence of a leak around the ETT. Temperature differences in degrees celsius will be reported.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: temperature difference degrees celsius
Arm/Group | Cuff Inflation and Cuff Deflation Groups
Number analyzed (Participants) | 50
temperature difference degrees celsius | 0.10 [0.04 to 0.16]

2. Secondary Outcome: Temperature Difference in the Presence of a Small Leak (Fractional Volume Loss < 21%) and Large Leak (Fractional Volume Loss > 21%)
Description: Sub-group analysis: Fractional Volume Loss (FVL) will be determined using spirometry readings taken during temperature measurements.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cuff Inflation and Cuff Deflation Groups
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 3/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cuff Inflation and Cuff Deflation Groups (N=59)
Nosebleed (Blood and lymphatic system disorders) | 1 — On insertion of nasopharyngeal temperature probe. Minor and self-resolved
Post-extubation stridor (Respiratory, thoracic and mediastinal disorders) | 1 — Self-resolved without medical therapy. Associated with use of Microcuff endotracheal tube
Partially obstructed ETT during emergence (Respiratory, thoracic and mediastinal disorders) | 1 — Associated with use of Microcuff endotracheal tube. Required suctioning with suction catheter, thereafter no further complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-03-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02201628/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT02201628/ICF_001.pdf